CLINICAL TRIAL: NCT02600143
Title: Identification of Predictive Parameters for Colitis in Melanoma Patients Treated With Immunotherapy.
Acronym: COLIPI
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: METc 2012/085
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Melanoma; Colitis
Keywords: Melanoma; Colitis; Ipilimumab; Nivolumab; Pembrolizumab
MeSH Terms: conditions — Melanoma; Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Intestinal biopsies, whole blood samples, stool samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this trial is to identify biomarkers and genetic predisposition for the development of immune checkpoint related colitis.

DETAILED DESCRIPTION:
Immunotherapy with immune checkpoint-inhibitors is standard treatment for patients with melanoma. However, in about 15% of patients treated with Ipilimumab a grade 3-4 colitis will occur. In programmed cell death protein 1 (PD1) inhibitors colitis is also seen as adverse event, although less prominent. We want to find a good predictive biomarker to select patients that are prone to colitis.So far no test is available that might be predictive whether a patient will develop a grade 3-4 colitis.

The study will consists of four parts: 1.) to identify a genetic profile associated with ipilimumab-induced colitis, 2.) to identify predictive (serum or fecal) biomarkers for ipilimumab-induced colitis, 3.) to study the tissue of ipilimumab-induced colitis and 4) to study the role of the gut microbiome in the development of colitis. Patients are able to participate in one, or more parts of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with melanoma who will be treated with immune checkpoint inhibitors (ipilimumab, nivolumab, pembrolizumab)
2. Signed written informed consent.
3. Able to comply with the protocol.

Exclusion Criteria:

1. Patients with a pre-existing colitis (e.g. Crohn's disease, ulcerative colitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2013-08; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Genetic predisposition for immunotherapy-induced colitis | 1 week
  Difference in genetic profile on 99 confirmed inflammatory bowel disease (IBD) loci between patients who develop immunotherapy-induced colitis and who do not.

SECONDARY OUTCOMES:
Predictive biomarkers for immunotherapy-induced colitis in stool and serum | Day 0, 21, 42, 63
  Comparison of calprotectin levels in the stool and serum-levels of C reactive protein (CRP), endotoxin, citrulline, intestinal fatty acid-binding protein (I-FABP), calprotectin and interleukin 8 (IL8) between patients who develop immunotherapy-induced colitis and who do not.
Clinical scoring system of colitis | Day -7 to 85
  Prediction of (severity of) colitis based on symptomatology measured with the MAYO score and BRISTOL stool scale.
Histological assessment of colon biopsies in patients that develop colitis | 1 day
  Immunotherapy-induced colitis will be assessed in colon biopsies when a sigmoidoscopy has to be performed for diagnostic reasons.
Analysis of the gut microbiome in stool samples | Day 0, 21, 42, 63
  Microbiome analysis in stool collected before treatment and at 3, 6, and 9 weeks and correlation with development of immunotherapy-induced colitis.

CONTACTS AND LOCATIONS:
Overall Officials: G. A.P. Hospers, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands